CLINICAL TRIAL: NCT03281070
Title: The Incidence and Risk Factors of Anastomotic Leakage After Anterior Resection of Rectal Cancer: a Multi-site Observational Study
Brief Title: Anastomotic Leakage After Anterior Resection of Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Department of General Surgery, Beijing Friendship Hospital
Other Study IDs: CR-AL
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-09

CONDITIONS: Rectal Cancer
Keywords: Anastomotic leakage; Anterior resection; Risk factors; Incidence; Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anastomotic leakage (AL) is one of the most-feared postoperative complications after anterior resection of rectal cancer. This complication compromises both short term and long term outcome of patients. The incidence of AL after anterior resection was approximately 6-11%. Although several risk factors for AL such as male sex, smoking, tumor location, longer operative time, intraoperative blood loss had been reported in previous studies, the incidence of AL did not meet a significant decrease. So far there is no multi-site observational study on incidence and risk factors of AL after anterior resection in China, therefore this study aims to work on this issue and provide evidence for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of the rectum by biopsy
* single lesion
* anterior resection was performed
* anastomosis using circular stapler

Exclusion Criteria:

* history of colorectal cancer surgery
* emergency surgery because of bowel obstruction, bleeding or perforation
* colo-anal anastomosis
* subtotal colectomy
* total colectomy
* abdominal perineal resection
* Hartmann procedure
* pull out anastomosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rectal cancer patients who underwent anterior resection with or without postoperative anastomotic leakage
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage | 14 days after surgery
  Anastomotic leakage is defined as a defect of the intestinal wall integrity at the colorectal anastomotic site leading to a communication between the intra- and extraluminal compartments.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China